CLINICAL TRIAL: NCT02970162
Title: A Phase 3, Double-Blind, Placebo-controlled, Randomized, Parallel-Group Study to Evaluate the Efficacy and Safety of Amifampridine Phosphate in Patients With Lambert-Eaton Myasthenic Syndrome
Brief Title: Phase 3 Study to Evaluate Efficacy of Amifampridine Phosphate in Lambert-Eaton Myasthenic Syndrome (LEMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMS-003
Expanded Access: NCT02189720 (Approved for marketing)
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Lambert-Eaton Myasthenic Syndrome
Keywords: LEMS
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- amifampridine phosphate (Experimental): amifampridine phosphate 10 mg (amifampridine equivalent) by mouth, 30 to 80 mg total daily dose, 3 to 4 times per day for 4 days
  Interventions: Drug: Amifampridine Phosphate
- placebo (for amifampridine phosphate) (Placebo Comparator): placebo by mouth 3 to 4 times per day for 4 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Amifampridine Phosphate
  Arms: amifampridine phosphate
Drug: Placebo Oral Tablet
  Arms: placebo (for amifampridine phosphate)

SUMMARY:
This study evaluates the effect of withdrawing amifampridine phosphate treatment from patients with LEMS. One half of the patients will continue to receive amifampridine phosphate and the other half will receive placebo, during this double-blind study.

DETAILED DESCRIPTION:
This was a randomized (1:1), double-blind, placebo-controlled, parallel-group, withdrawal study designed to evaluate the efficacy and safety of amifampridine phosphate in patients diagnosed with LEMS. The study was planned to include approximately 28 male and female patients.

Prior to the study, patients were receiving unblinded treatment in the expanded access program (EAP-001). Patients had to be on a stable dose and frequency of amifampridine phosphate for at least 1 week prior to randomization into LMS-003. Screening and randomization (Day 0) may have been into a single visit.

Patients who met eligibility criteria were randomized 1:1 to amifampridine phosphate (at the patient's optimal dose) or placebo on Day 0.

Baseline assessments were obtained on Study Day 0, while the patient has been on open-label amifampridine phosphate and in relationship to the usual dosing schedule. Patients took blinded study medication on Day 1 through Day 3. On Day 4, a dose of blinded study medication was administered by the site study personnel. This was the same medication that the patient took on Day 1 through Day 3. The assessments listed below were performed following either the second, third, or fourth dose of medication taken on Day 4, and this should be the same dose after which Day 0 assessments were performed. For example, if the patient took their second dose of amifampridine in the clinic on Day 0 and had assessments started 40 minutes later, then on Day 4, that patient should be assessed after taking their second dose of investigational product (IP).

Beginning with the next dose after all Day 0 baseline assessments were completed, the patient received IP through Day 4, with a clinic visit on the last day (Day 4) for assessments.

The planned duration of participation for each patient was up to 12 days, including screening (up to 7 days), Day 0 assessments and randomization, and IP administration (Day 1 through Day 4).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age and currently receiving amifampridine phosphate for LEMS.
2. Diagnosis of LEMS by antibody testing or electromyography (EMG).
3. Completion of anti-cancer treatment at least 3 months (90 days) prior to Screening.
4. If receiving peripherally acting cholinesterase inhibitors (e.g. pyridostigmine), a stable dose of cholinesterase inhibitors is required for at least 7 days prior to randomization and throughout the study.
5. If receiving permitted oral immunosuppressants (prednisone or other corticosteroid), a stable dose is required for at least 30 days prior to randomization and throughout the study.
6. Female patients of childbearing potential must practice an effective, reliable contraceptive regimen during the study.
7. Able to perform all study procedures and assessments.
8. Willing and able to travel to study site and attend all clinic study visits.
9. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Clinically significant long corrected QT (QTc) interval on ECG in previous 12 months.
2. Seizure disorder.
3. Active brain metastases.
4. Unable to ambulate.
5. Pregnant or lactating females.
6. Any other condition which, in the opinion of the Investigator, might interfere with the patient's participation in the study or confound the assessment of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Shieh, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Amifampridine Phosphate: amifampridine phosphate 10 mg (amifampridine equivalent) by mouth, 30 to 80 mg total daily dose, 3 to 4 times per day for 4 days
  Amifampridine Phosphate
- Placebo (for Amifampridine Phosphate): placebo by mouth 3 to 4 times per day for 4 days
  Placebo Oral Tablet
Period: Overall Study
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.51) | 53.4 (13.46) | 54.2 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 77.62 (20.312) | 93.95 (15.449) | 85.78 (19.545)

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Myasthenia Gravis (QMG) Score
Description: The QMG is a physician-rated test including 13 assessments such as facial strength, swallowing, grip strength, and duration of time that limbs can be maintained in outstretched positions. Each assessment is graded as 0 (none), 1 (mild), 2 (moderate), or 3 (severe), for a total range of 0-39. A higher total score indicates a worse outcome.
Time Frame: change from baseline in QMG score at end of day 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate)
Number analyzed (Participants) | 13 | 13
scores on a scale
  Baseline | 7.8 (4.20) | 8.5 (5.43)
  Day 4 | 7.9 (4.94) | 15.0 (5.90)
  Change from baseline | 0.1 (3.07) | 6.5 (4.82)
Statistical Analysis 1: Comparison: Amifampridine Phosphate vs Placebo (for Amifampridine Phosphate); Test type: Superiority; p = 0.0004, Least square means — LS means; Fixed effects treatment and QMG at Baseline. Between-treatment difference in LS means (95% CI) -6.54 (-9.78, -3.29)

2. Primary Outcome: Subject Global Impression (SGI) Score
Description: The SGI is a 7-point scale on which the patient rates their global impression of the effects of a study treatment (1=terrible to 7=delighted). The SGI was assessed by the patient or the patient's parent/guardian/caregiver if the patient was unable to complete the SGI. The SGI has demonstrated concordance with the physician's assessment of improvement.
Time Frame: change from baseline in SGI score at end of day 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate)
Number analyzed (Participants) | 13 | 13
scores on a scale
  Baseline | 6.1 (0.86) | 5.8 (0.90)
  Day 4 | 5.3 (1.65) | 2.4 (1.76)
  Change from baseline to Day 4 | -0.8 (1.74) | -3.5 (2.18)
Statistical Analysis 1: Comparison: Amifampridine Phosphate vs Placebo (for Amifampridine Phosphate); Test type: Superiority; p = 0.0003, Fixed effects linear model — CFB for SGI score was modeled as the response, with fixed effects terms for treatment and SGI at Baseline; This statistical test applies to the change from baseline SGI scores to Day 4 values row; LS means = 2.95, 95% CI 2-sided [1.53 to 4.38]

3. Secondary Outcome: Change in Clinician's Global Impression of Improvement (CGI-I) at Day 4 Compared to Baseline
Description: The CGI-I captures the Investigator's global impression of the patient's improvement or worsening from baseline status. The 7-point scale is scored by the Investigator based on changes in symptoms, behavior, and functional abilities. Each symptom is rated as 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), or 7 (very much worse). The total score can range from 0 to 49. A higher score indicates a worse outcome.
Time Frame: change from baseline in CGI-I score at end of day 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate)
Number analyzed (Participants) | 13 | 13
scores on a scale | 3.8 (0.8) | 5.5 (1.27)
Statistical Analysis 1: Comparison: Amifampridine Phosphate vs Placebo (for Amifampridine Phosphate); Test type: Superiority; p = 0.0020, Wilcoxon Rank Sum Test

4. Other Pre Specified Outcome: Triple Timed Up and Go Walk Test (3TUG)
Description: The 3TUG is a functional mobility test that requires a patient to stand up from a straight-backed armchair, walk 3 meters, turn around, walk back, and sit down in the chair. A modification of this is where the individual performs the test 3 times without pause, and the measurement is the average time required to complete each of the 3 repetitions. Based upon literature reports that a significant change in gait for a similar walk-test is an increase in time of more than 20%, this has been incorporated into the endpoint.
Time Frame: change from baseline in 3TUG at end of day 4
Population: The number and proportion of patients with a ≥20% increase in 3TUG average time
Measure: Count of Participants; unit: Participants
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate)
Number analyzed (Participants) | 13 | 13
Participants | 1 | 8
Statistical Analysis 1: Comparison: Amifampridine Phosphate vs Placebo (for Amifampridine Phosphate); Test type: Superiority; p = 0.0112, Fisher Exact

ADVERSE EVENTS:
Time Frame: All AEs were observed for each patient from enrollment until study completion (up to 12 days per patient).
Description: Treatment-emergent AEs (TEAEs) were summarized using system organ class and PT by treatment and overall for all patients in the safety population.
Arm/Group | Amifampridine Phosphate | Placebo (for Amifampridine Phosphate)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amifampridine Phosphate (N=13) | Placebo (for Amifampridine Phosphate) (N=13)
atrial fibrillation (Cardiac disorders) | 0 | 1
myocardial ischemia (Cardiac disorders) | 0 | 4
motion sickness (Ear and labyrinth disorders) | 0 | 1
diplopia (Eye disorders) | 0 | 1
eyelid ptosis (Eye disorders) | 0 | 1
dry mouth (Gastrointestinal disorders) | 0 | 2
diarrhoea (Gastrointestinal disorders) | 0 | 1
dysphagia (Gastrointestinal disorders) | 0 | 1
hypoaesthesia, oral (Gastrointestinal disorders) | 0 | 1
impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 0 | 1
oral disorder (Gastrointestinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
fatigue (General disorders) | 0 | 4
asthenia (Gastrointestinal disorders) | 0 | 2
feeling hot (General disorders) | 0 | 2
gait disturbance (General disorders) | 0 | 1
pain (General disorders) | 0 | 1
bronchitis (Infections and infestations) | 0 | 1
decreased appetite (Metabolism and nutrition disorders) | 0 | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5
limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
balance disorder (Nervous system disorders) | 0 | 2
eyelid ptosis (Nervous system disorders) | 0 | 1
facial nerve disorder (Nervous system disorders) | 0 | 1
headache (Nervous system disorders) | 1 | 0
movement disorder (Nervous system disorders) | 0 | 1
somnolence (Nervous system disorders) | 0 | 1
speech disorder (Nervous system disorders) | 0 | 1
insomnia (Psychiatric disorders) | 0 | 1
dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT02970162/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02970162/SAP_001.pdf